CLINICAL TRIAL: NCT05340283
Title: Clinical-epidemiological Characteristics of Patients With Parkinson's Disease Referred to a Home Rehabilitation Service
Brief Title: Parkinson's Disease in Home Rehabilitation Services
Status: Completed | Type: Observational
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, María Cruz Sousa Fraguas, Principal investigator: Physiotherapist., University of Oviedo
Other Study IDs: 243-2021 Parkinson´s disease
Record Dates: First submitted 2022-04-12; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Parkinsonian disorders; Home care services; Home care agencies; Rehabilitation; Physical therapy modalities
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational group: Patients with Parkinson's disease who were referred to a Home Rehabilitation Service in Gijón, Asturias region, Spain, during the years 2015 to 2021.
  Interventions: Procedure: physiotherapy

INTERVENTIONS:
Procedure: physiotherapy — Patients received physiotherapy treatment at home for a certain period of time. Data were collected on the assessments made at the beginning and at the end of the physiotherapy treatment.
  Other Names: Physiotherapy treatment

SUMMARY:
Introduction: Home rehabilitation is a form of care that is part of most health systems. Patients with Parkinson's disease can be referred to these Home Rehabilitation Services given the characteristics of the pathology they suffer.

Objective: know and analyse the clinical-epidemiological characteristics of patients with Parkinson's disease referred to a Home Rehabilitation Service belonging to health Area V of Gijón, Asturias, Spain.

Study Design: This project proposes an observational and retrospective study.

Study population: The subjects that will be part of this study will be men and women with Parkinson's disease who have been referred to the Home Rehabilitation Service from 2015 to 2021.

DETAILED DESCRIPTION:
Introduction:

Home-based rehabilitation is a care modality that is part of most healthcare systems. In most cases, patients are referred from hospitals, by the rehabilitation services themselves or by the specialist physicians who have treated them. Patients who may be candidates for home rehabilitation often have difficulties in accessing a hospital or outpatient centre independently, due to difficulty in walking and/or architectural barriers within or outside the home, so that in order to travel to outpatient centres, they need means of transport such as ambulances, which entails high costs. Patients with Parkinson's Disease can be referred to these Home Rehabilitation Services.

Objectives:

General:

Know and analyse the clinical-epidemiological characteristics of patients with Parkinson's Disease referred to a Home Rehabilitation Service belonging to the Health Area V of Gijón.

Specific:

Assess the distribution of patients by age group, sex, social conditions and degree of functional impairment.

Find out the time needed for recovery or completion of treatment, as well as the criteria for discharge.

Obtain information on the social assessment and architectural barriers of Parkinson's disease patients referred to a Home Rehabilitation Service.

Study design:

The present project proposes to carry out an observational, ex post facto, retrospective study.

The subjects who will be part of this study will be men and women with Parkinson's disease who have been referred to the Home Rehabilitation Service from 2015 to 2021. Available data from the entire population of patients with Parkinson's disease who meet the inclusion criteria will be analysed.

Limitations:

The limitations of the present study are that the patients will be analysed within a specific setting, such as a Home Rehabilitation Service, so it is possible that some results cannot be generalized.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with Parkinson's disease
* Patients belonging to Health Area V of the Health System of the Principality of Asturias, Spain.
* Subjects who have been referred at some point to home rehabilitation.

Exclusion Criteria:

- Patients who have been discharged at the first medical visit.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Diagnosis: | Baseline
  The specific diagnosis of Parkinsonian syndrome presented by each patient.
Epidemiological characteristics | Baseline
  Age, this variable will be measured in years. Sex will be recorded as male and female. Social assessment: the following data will be recorded: Place of residence: whether the patient lives alone at home, with his or her family or in a geriatric centre. Existence or non-existence of a caregiver, if so, whether it is formal or informal. Housing suitable for the patient's needs or not. Finally, comorbidities: according to the Charlson comorbidity index, considering absence of comorbidity between 0 and 1 points, low comorbidity 2 points, high comorbidity between 3 and 5 points and severe comorbidity over 5 points.

SECONDARY OUTCOMES:
Barthel index | Baseline to end of treatment (up to 3 months)
  Functional independence was measured by the Barthel Index. It has a total score ranging from 0 to 100, where 0 is the minimum (worst outcome) and 100 is the maximum (best outcome).
Pain intensity | Baseline to end of treatment (up to 3 months)
  Numerical visual analogue pain measurement scale. The patient must assign a numerical value to the pain between two extreme points (0 no pain, to 10 the worst pain imaginable), the higher the score the greater the pain experienced.
Gait assessment | Baseline to end of treatment (up to 3 months)
  Gait ability measured according to Holden's Gait Classification (FAC). This scale ranges from 0 (no gait) to 5 (independent gait including walking up and down stairs). The higher the score, the better the gait performance.
Reason for discharge | End of treatment (up to 3 months)
  Can be the following options:
  * The value of the Barthel index reached at the end of treatment.
  * Chronicity.
  * Referral to outpatient rehabilitation.
  * Change of residence.
  * Voluntary discharge.
  * Hospital admission.
  * Worsening without hospital admission.
  * Exitus.

CONTACTS AND LOCATIONS:
Overall Officials: María Cruz Sousa-Fraguas, Principal Investigator — University of Oviedo